CLINICAL TRIAL: NCT05783323
Title: Larotrectinib to Enhance RAI Avidity in Patients With Differentiated Thyroid Cancer Harboring NTRK Fusions (LANTERN)
Brief Title: Larotrectinib to Enhance RAI Avidity in Differentiated Thyroid Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-020549
Record Dates: First submitted 2023-03-02; First posted 2023-03-24 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Differentiated Thyroid Cancer; Pediatric Cancer; Cancer; Cancer, Thyroid
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be an open label, non-randomized study to evaluate the efficacy and safety of the combination of larotrectinib followed by 131I therapy for patients with NTRK fusion differentiated thyroid cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Larotrectinib monotherapy with 131I therapy (Experimental): Patients will receive larotrectinib monotherapy for 6 months at the FDA-approved dose.
  Patients will receive 131I therapy after 6 months of larotrectinib. Larotrectinib will be continued for 5 days after RAI therapy and then patients will enter a wait and see period off treatment.
  Patients who experience disease progression at any point while on larotrectinib will proceed to 131I therapy and discontinue larotrectinib.
  Interventions: Drug: Larotrectinib monotherapy; Radiation: 131I therapy

INTERVENTIONS:
Drug: Larotrectinib monotherapy — Patients will receive larotrectinib monotherapy for 6 months at the FDA-approved dose.
Radiation: 131I therapy — Patients will receive 131I therapy after 6 months of larotrectinib.

SUMMARY:
Papillary thyroid cancer (PTC) is the most common form of differentiated thyroid cancer (DTC). The traditional first line treatment for patients with advanced DTC after surgical resection is radioactive iodine (RAI) therapy. However, less than a quarter of patients with lung metastases will achieve a complete response to RAI therapy, and this therapy carries the risk of pulmonary fibrosis and an increasingly recognized risk of secondary malignancies.

DETAILED DESCRIPTION:
This is an open label, non-randomized study to evaluate the efficacy and safety of the combination of larotrectinib followed by 131I therapy for patients with NTRK fusion differentiated thyroid cancer. The primary Phase II objective will be to evaluate the pulmonary structural response rate at 18 months to the combination of larotrectinib given for 6-months followed by 131I therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 1 year
2. Histologic diagnosis of a differentiated thyroid cancer, s/p thyroidectomy and adequate local therapy (e.g., lymph node dissection as per standard of care) for metastatic disease in the neck in the opinion of the treating investigator
3. Anatomically evaluable disease on chest CT meeting one of the following criteria (obtained within 90 days of enrollment):

   A. multiple (> 10) noncalcified solid pulmonary nodules visible on CT and/or B. enlarging, discrete pulmonary nodules visible on CT of any number consistent with metastatic disease
4. Identification of an neurotrophic tyrosine receptor kinase (NTRK) (NTRK1, NTRK2, or NTRK3) gene fusion in a CLIA/CAP accredited laboratory without known kinase domain resistance mutation
5. Lansky/Karnofsky performance status ≥ 50%
6. Adequate Organ Function

   A. Bone Marrow Function:
   * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3
   * Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   * Hemoglobin ≥ to 8.0 g/dL at baseline (may receive red blood cell (RBC) transfusions).

   B. Adequate Renal Function:

   Creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m2 or a maximum serum creatinine based on age/gender as follows:

   Age Maximum Serum Creatinine (mg/dL) Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.5

   ≥ 16 years 1.7 1.7

   C. Adequate Liver Function
   * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age.
   * Serum glutamic-pyruvic transaminase (SGPT) (ALT) ≤ 135 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
   * Serum albumin ≥ 2 g/dL
7. Female patients of reproductive potential must agree to use a highly effective contraceptive method for the duration of study therapy and for at least one month after the final dose of larotrectinib. Males of reproductive potential with a non-pregnant female partner of child-bearing potential must use a highly effective contraception for the duration of the study and for at least one month after the final dose of larotrectinib.

Exclusion Criteria

1. No prior systemic therapy for thyroid cancer, including tropomyosin receptor kinase (TRK) inhibitors. Note that prior 131I is permitted.
2. Females who are pregnant or breastfeeding are excluded due to the potential risks of larotrectinib and RAI to the fetus/neonate.
3. Concurrent therapy: Patients currently receiving a strong CYP3A4 inducer or inhibitor are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided 14 days prior to treatment to the end of the study treatment.

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete pulmonary structural response | 18 months
  The primary endpoint is the complete pulmonary structural response rate to larotrectinib by modified Nies et al thyroid cancer response criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Laetsch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No